CLINICAL TRIAL: NCT06837103
Title: Real-world Effects of Using Intermittently Scanned Continuous Glucose Monitoring and Pharmacist-led Coaching on the Management of Type 2 Diabetes Among Adults Using Non-insulin Antihyperglycemic Agents
Brief Title: Real-world Effects of Using Intermittently Scanned Continuous Glucose Monitoring and Pharmacist-led Coaching on the Management of Type 2 Diabetes Among Adults Not Using Insulin (REAL isCGM T2D)
Acronym: REAL isCGM T2D
Status: Recruiting | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Sun Life Assurance Company of Canada (Unknown)
Responsible Party: Sponsor
Other Study IDs: REAL isCGM T2D
Record Dates: First submitted 2025-01-29; First posted 2025-02-20 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: continuous glucose monitoring; type 2 diabetes; time in range; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- isCGM Group: Adults with T2D, who are active patients at LMC, not using insulin, and initiate a second generation isCGM device through Lumino Health™ Pharmacy, and complete one initial pharmacist consultation
  Interventions: Device: Intermittently Scanned Continuous Glucose Monitor
- CBG Group: Adults with T2D, who are active patients at LMC, not using insulin and use a CBG monitor
- isCGM+Coaching Group: Adults with T2D, who are active patients at LMC, not using insulin, and initiate a second generation isCGM device through Lumino Health™ Pharmacy, and complete 2 or more diabetes coaching program consultations
  Interventions: Device: Intermittently Scanned Continuous Glucose Monitor

INTERVENTIONS:
Device: Intermittently Scanned Continuous Glucose Monitor — intervention used by the isCGM and isCGM+Coaching groups
  Groups: isCGM Group; isCGM+Coaching Group

SUMMARY:
The goal of this prospective study is to evaluate diabetes outcomes after initiating second generation intermittently scanned continuous glucose monitoring (isCGM) plus one pharmacist consultation session compared with capillary blood glucose (CBG) monitoring among insulin-naïve adults with type 2 diabetes (T2D) in a specialist endocrinology clinical setting in Canada.

Primary Outcome - To evaluate change in HbA1c at 3-6 months follow-up after initiating isCGM plus one pharmacist consultation (isCGM cohort) compared with CBG monitoring (CBG cohort) among insulin-naïve adults with T2D.

Secondary Outcomes - To determine the change in metabolic outcomes and patient reported outcomes (PROs) and number of non-insulin antihyperglycemic agents (AHAs) prescribed from baseline to 3-6 months (± 6 weeks) in the isCGM cohort compared to the CBG cohort. Another secondary outcome is to assess isCGM metrics and number of isCGM discontinuations in the isCGM cohort at 3-6 months (± 6 weeks) compared to baseline. Additionally the study will describe and/or evaluate glycemic and metabolic outcomes, and PROs in participants who initiate an isCGM device and opt to enroll in a diabetes coaching program (isCGM+coaching cohort) at baseline compared to follow-up at 3-6 months (± 6 weeks).

Exploratory Outcomes - To compare change in HbA1c between the matched isCGM cohort and CBG cohort by subgroups: age (< 65 years old vs ≥ 65 years old) and baseline HbA1c (< 8.5% vs ≥ 8.5%).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Clinical diagnosis of T2D ≥ one year
* Using at least one AHA
* Status as a Sun Life group benefits member, initiates isCGM device through Lumino Health™ Pharmacy, and completes one initial pharmacist consultation (isCGM cohort) or completes 2 or more diabetes coaching program consultations (isCGM+coaching cohort); or has private health insurance and uses CBG monitoring (CBG cohort)
* Baseline HbA1c ≥ 7.0%
* ≥ 1 HbA1c value up to 6 months prior to index date
* Exclusive use of isCGM for ≥ 3 months
* Informed consent

Exclusion Criteria:

* Have a history of insulin use
* Are pregnant or breastfeeding at the time of study enrollment or become pregnant during the study
* Have an estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2
* Previously used rtCGM or isCGM for > 3 months
* Recent or expectant change to antihyperglycemic medications or doses within 30 days of index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adults with T2D, who are active patients at LMC, not using insulin, and initiate a second generation isCGM device through Lumino Health™ Pharmacy, and complete one initial pharmacist consultation (isCGM cohort) or complete 2 or more diabetes coaching program consultations (isCGM+coaching cohort), or use a CBG monitor (CBG cohort)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | from enrollment to 3-6 month follow up
  Evaluate the change in HbA1c at 3-6 months follow-up (±6 weeks) in the matched isCGM and CBG cohorts among adults with insulin-naïve T2D

SECONDARY OUTCOMES:
Change in Weight | from enrollment to 3-6 month follow up
  Evaluate the change in weight in the isCGM and CBG cohorts
Change in BMI | from enrollment to 3-6 month follow up
  Evaluate the change in body mass index (BMI) in the isCGM and CBG cohorts
Change in Blood Pressure | from enrollment to 3-6 month follow up
  Evaluate the change in blood pressure in the isCGM and CBG cohorts
Proportion of Participants Achieving HbA1c ≤ 7.0% at Follow-Up | from enrollment to 3-6 month follow up
  Evaluate the proportion of participants achieving HbA1c ≤ 7.0% at follow-up in the isCGM and CBG cohort
Proportion of Participants with ≥1 Self-Reported Hypoglycemic Event per Week | from enrollment to 3-6 month follow up
  Evaluate the proportion of participants with ≥1 self-reported hypoglycemic event per week in the isCGM and CBG cohort
Percent Time in Range (TIR) | from enrollment to 3-6 month follow up
  Evaluate percent time in range (3.9 to 10.0 mmol/L) in the isCGM and isCGM+Coaching cohorts
Percent Time Below Range (TBR) | from enrollment to 3-6 month follow up
  Evaluate percent time below range (< 3.9 mmol/L) in the isCGM and isCGM+Coaching cohorts
Percent Time Below Range (TBR) in Level 2 Hypoglycemia | from enrollment to 3-6 month follow up
  Evaluate Percent TBR in level 2 hypoglycemia (< 3.0 mmol/L) in the isCGM and isCGM+Coaching cohorts
Percent Time Above Range (TAR) | from enrollment to 3-6 month follow up
  Evaluate Percent TAR (> 10.0 mmol/L) in the isCGM and isCGM+Coaching cohorts
Estimated Glucose Management Indicator (eGMI) | from enrollment to 3-6 month follow up
  Evaluate the Estimated Glucose Management Indicator (eGMI) in the isCGM and isCGM+Coaching cohorts
Mean glucose | from enrollment to 3-6 month follow up
  Evaluate mean glucose in the isCGM and isCGM+Coaching cohorts
Glycemic variability | from enrollment to 3-6 month follow up
  Evaluate glycemic variability reported as SD and CV in the isCGM and isCGM+Coaching cohorts
Percent sensor capture | from enrollment to 3-6 month follow up
  Evaluate percent sensor capture in the isCGM and isCGM+Coaching cohorts
Number of isCGM discontinuations | assessed at 3-6 month follow-up
  Evaluate the number of isCGM discontinuations in the isCGM and isCGM+Coaching cohorts only at follow-up
Number of diabetes coaching program discontinuations | from enrollment to 3-6 month follow up
  Evaluate the number of diabetes coaching program discontinuations, measured by the Diabetes Coaching Program survey in the isCGM and isCGM+Coaching cohorts
Psychological distress | from enrollment to 3-6 month follow up
  Evaluate psychological distress measured by the Diabetes Distress Scale (DDS) in the isCGM and isCGM+Coaching cohorts
Glucose monitoring device satisfaction | from enrollment to 3-6 month follow up
  Evaluate glucose monitoring device satisfaction measured by the Glucose Monitoring System Satisfaction Scale (GMSS) in the isCGM and isCGM+Coaching cohorts
Proportion of participants achieving HbA1c ≤ 7.0% | assessed at 3-6 month follow-up
  Evaluate proportion of participants achieving HbA1c ≤ 7.0% in the isCGM and isCGM+Coaching cohorts at follow-up only
Change in Weight | from enrollment to 3-6 month follow up
  Evaluate change in weight in only the isCGM+Coaching cohort
Change in Body Mass Index (BMI) | from enrollment to 3-6 month follow up
  Evaluate the change in body mass index in only the isCGM+Coaching cohort
Change in Blood Pressure | from enrollment to 3-6 month follow up
  Evaluate Change in Blood Pressure in only the isCGM+Coaching cohort
Proportion of participants with ≥1 self-reported hypoglycemic event per week | from enrollment to 3-6 month follow up
  Evaluate the proportion of participants with ≥1 self-reported hypoglycemic event per week in the isCGM+Coaching cohort only

OTHER OUTCOMES:
Change in HbA1c by Age | assessed at 3-6 month follow-up
  Evaluate change in HbA1c at 3-6 months follow-up (±6 weeks) in the matched isCGM and CBG cohorts among adults with insulin-naïve T2D by age < 65 years old vs ≥ 65 years old subgroups
Change in HbA1c by Baseline HbA1c | assessed at 3-6 month follow-up
  Evaluate change in HbA1c at 3-6 months follow-up (±6 weeks) in the matched isCGM and CBG cohorts among adults with insulin-naïve T2D by baseline HbA1c (< 8.5% vs ≥ 8.5% subgroups)

CONTACTS AND LOCATIONS:
Locations (1):
- LMC Diabetes & Endocrinology Ltd., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a real-world study using data from a national Diabetes Registry. IPD will not be shared.